CLINICAL TRIAL: NCT06588881
Title: A Pilot Study on Feasibility of Technique, Performance and Safety of ENDONEB Endoscopic Medical Device for the Nebulized Application of the Haemostatic Surgical Sealant After Gastrointestinal Endoscopic Resection
Brief Title: Endoscopic Nebulizing Device for Surgical Haemostatic-sealant Glubran® 2 Usability Trial in EMR and ESD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GEM SRL (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: DGDMF/I.5.i.m.2/2022/2045
Record Dates: First submitted 2024-08-07; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Intervention Model Description: Single center, prospective, medical device usability and feasibility study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ENDONEB (Other): The sterile device and gamma rays, latex free and disposable consists of the following components: a steel canister, a catheter 2m hose, one attack base located at the proximal end of the catheter, one unit at the end back, two needles and two syringes. The device must always be stored in the original packaging. Store only in one place Temp temperature not exceeding 30°C(86°)Application procedure: The device must be pr repaired and activated adequately in order to ensure its correctness operation. See instructions for assembly and indoor use of the package.
  Interventions: Device: nebulized application of the haemostatic surgical sealant after gastrointestinal endoscopic resection

INTERVENTIONS:
Device: nebulized application of the haemostatic surgical sealant after gastrointestinal endoscopic resection — ENDONEB, a nebulizing catheter containing the synthetic haemostatic-sealant Glubran®, is inserted in the operative channel of the endoscope until it is pushed out of the endoscope tip approximately 2 cm. The haemostatic-sealant is nebulized over the surface of the post resection mucosal defect by activating the propellant (medical-inert-gas) container. An amount of about 0.3 mL of Glubran® 2 (or more - depending on dimension of the lesion) is applied on mucosal or sub-mucosal defect in order to create a proper haemostaticsealant film.

SUMMARY:
The aim of this single-center study is to evaluate the feasibility of the technique, usability and safety of the device ENDONEB.

DETAILED DESCRIPTION:
Single center, prospective, medical device usability and feasibility study. The study will be performed in Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome.

According to the recomandations of the Italian Ministry of Health (28) regarding the sample size of pilot and feasibility studies, 15 applications underwent to mucosal or submucosal resection procedures will be evaluated. The recruitment period will be 36 weeks (9 months). The evaluation ends when ENDONEB has been used in the fifteenth subject or at one third of applications if the investigators will be able to give their evaluation of the feasibility of the ENDONEB technique, usability and safety. The ENDONEB medical device belongs to the family of "Nebulizers" class IIa accessory devices, used to apply Glubran®2 in nebulized form in laparotomic, laparoscopic and thoracoscopic procedures. The ENDONEB medical device allows to apply the Glubran®2 in nebulized form in digestive endoscopy interventions and can be used both with gastroscopes and colonoscopes with an operating channel not less than 2.6 mm. It is marketed in sterile presentation; the components are latex free and is for single use only.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of superficial neoplastic lesion to be resected by a gastrointestinal endoscopic resection (EMR or ESD)
* Older than 18 years of age at time of consent;
* Operable per institution's standards;
* Signed and dated informed consent form

Exclusion Criteria:

* Any clinical conditions precluding the feasibility of gastrointestinal endoscopic resection (ENDONEB could be contraindicated in patients who are suspected of having a gastrointestinal perforation, or are at high risk of gastrointestinal perforation during endoscopic treatment);
* Pregnant during period of study participation;
* Allergy history to cyanoacrylate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Evaluate the feasibility of the technique | From the beginning of the surgery until the end of surgery. Approximately 3 hours.
  Appropriateness of ENDONEB medical nebulizer device to apply the surgical haemostatic-sealant Glubran® 2 after gastrointestinal endoscopic resections evaluated in terms of positioning correctly the ENDONEB device for procedure as per the user manual's instructions. The outcome is measured with score 1-5 corresponding to the quality assessment: 1=not sufficient; 2=sufficient; 3=good; 4=very good; 5=excellent.
Evaluate the feasibility of the technique | From the beginning of the surgery until the end of surgery. Approximately 3 hours.
  Appropriateness of ENDONEB medical nebulizer device to apply the surgical haemostatic-sealant Glubran® 2 after gastrointestinal endoscopic resections evaluated in terms of facility of use and satisfaction/effectiveness of the surgeon. The outcome is mesaured with score 1-5 corresponding to the quality assessment: 1=not sufficient; 2=sufficient; 3=good; 4=very good; 5=excellent.

SECONDARY OUTCOMES:
Evaluate the ENDONEB Usability and Safety | From the beginning of the surgery until the end of surgery. Approximately 3 hours.
  Performance: evaluation of the device under anticipated conditions of use will be get by testing (verifying) the following issues:
  • the facility to assembly the device (setting up time, easiness in assembly, single operator assembly). Each point is mesaured with score 1-5 corresponding to the quality assessment: 1=not sufficient; 2=sufficient; 3=good; 4=very good; 5=excellent.
Evaluate the ENDONEB Usability and Safety | From the beginning of the surgery until the end of surgery. Approximately 3 hours.
  Performance: evaluation of the device under anticipated conditions of use will be get by testing (verifying) the following issues:
  • the ability to deliver the haemostatic-sealant to the resection site. The outcome is mesaured with score 1-5 corresponding to the quality assessment: 1=not sufficient; 2=sufficient; 3=good; 4=very good; 5=excellent.
Evaluate the ENDONEB Usability and Safety | From the beginning of the surgery until the end of surgery. Approximately 3 hours.
  Performance: evaluation of the device under anticipated conditions of use will be get by testing (verifying) the following issues:
  • the ability to use the device through the endoscope. The outcome is mesaured with score 1-5 corresponding to the quality assessment: 1=not sufficient; 2=sufficient; 3=good; 4=very good; 5=excellent.
Evaluate the ENDONEB Usability and Safety | From the beginning of the surgery until the end of surgery. Approximately 3 hours.
  Performance: evaluation of the device under anticipated conditions of use will be get by testing (verifying) the following issues:
  • the duration of the procedure to use the device (time). The outcome is mesaured in minutes.
Evaluate the ENDONEB Usability and Safety | From the beginning of the surgery until the end of surgery. Approximately 3 hours.
  Performance: evaluation of the device under anticipated conditions of use will be get by testing (verifying) the following issues:
  • ease of use in terms of capacity to control and manage the device. The outcome is mesaured with score 1-5 corresponding to the quality assessment: 1=not sufficient; 2=sufficient; 3=good; 4=very good; 5=excellent.
Evaluate the ENDONEB Usability and Safety | From the beginning of the surgery until the end of surgery. Approximately 3 hours.
  Performance: evaluation of the device under anticipated conditions of use will be get by testing (verifying) the following issues:
  • any technical complications during the procedure of application. The evaluation of this outcome is a detailed description of the technical complications that occurred.
Evaluate the ENDONEB Usability and Safety | From the beginning of the surgery until the end of surgery. Approximately 3 hours.
  Safety assessment will be performed by verifying any episodes of device malfunction during the entire application such as:
  • failure or breakage of the device. The measure of this outcome is reported with a detailed description of the event.
Evaluate the ENDONEB Usability and Safety | From the beginning of the surgery until the end of surgery. Approximately 3 hours.
  Safety assessment will be performed by verifying any episodes of device malfunction during the entire application such as:
  • lengthening of application times due to obstruction of the catheter or obstruction of the operating channel. The outcome is measured with a score from 1 to 5 corresponding to the quality assessment: 1=not sufficient; 2=sufficient; 3=good; 4=very good; 5=excellent.

CONTACTS AND LOCATIONS:
Overall Officials: Cristiano Spada, DR, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy, Italy